CLINICAL TRIAL: NCT06220136
Title: Comparison of the Performances of the Train-of-Four Ratio and the Modified Train-of-Four Ratio During Reversal of Deep Neuromuscular Blockade With Sugammadex
Brief Title: Comparison of the Performances of the cTOFR and the mTOFR During Reversal of Deep Neuromuscular Blockade With Sugammadex
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice Güneş Yeşilova, MD, Research assistant, Ankara University
Other Study IDs: 1357Hg*
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neuromuscular Blockade; Anesthesia, General
Keywords: neuromuscular blockade; neuromuscular junction monitoring; TOFscan; modified TOF ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single group: rocuronium drug administration TOFscan monitoring administration of sugammadex drug recording of classical TOF and modified TOF values
  Interventions: Device: TOFscan monitoring

INTERVENTIONS:
Device: TOFscan monitoring — observation and data recording

SUMMARY:
It is known that deep neuromuscular block improves surgical conditions, especially during laparoscopic abdominal surgery. Based on this, in the Perioperative Neuromuscular Blockade Management guide published by the ESAIC association in 2022, it is recommended to deepen the level of neuromuscular blockade in cases where surgical conditions need to be improved. Sugammadex should be used to quickly and reliably reverse deep neuromuscular blockade. TOFScan, a 3-dimensional acceleromyograph for neuromuscular monitoring, has become widely used in recent years. With this monitor, it has been shown that in addition to the classical train-of-four ratio (cTOFR), the modified train-of-four ratio (mTOFR) can be used during the spontaneous recovery of nondepolarizing neuromuscular blockade. In a study conducted by Schmartz et al. in 2021, it was shown that mTOFR, which is the ratio of T4 to the reference stimulus, was compiled later than cTOFR. Therefore, it is suggested that the mTOFR value is a better determinant for safe extubation.

DETAILED DESCRIPTION:
Neuromuscular blockers (NMB) agents are commonly used drugs in anesthesia for facilitating airway management, improving surgical conditions, and inducing immobility in critical situations. As a natural consequence of their use, postoperative residual neuromuscular block has been associated with serious postoperative complications such as upper airway obstruction, reintubation, atelectasis, pneumonia, prolonged stay in the post-anesthesia care unit (PACU), and decreased patient satisfaction. The incidence of residual block at the end of surgery and/or in the PACU is approximately 64% according to the literature .

Various factors contribute to the high incidence of residual neuromuscular block, including variability in the duration of action of neuromuscular blocker agents, variability in the time it takes for antagonist drugs to restore neuromuscular function, and clinicians' reliance on unreliable methods for assessing neuromuscular strength, such as continuous head lifting, grip strength, or respiratory measurements (e.g., tidal volume, inspiratory force), and the subjective evaluation of peripheral nerve stimulation responses . Residual neuromuscular block is a significant patient safety concern, and its detection and risk reduction are crucial for improving patient outcomes. One of the objective methods for assessing neuromuscular function is the Train of Four (TOF), which is an acceleromyographic peripheral nerve stimulator.

The effectiveness of TOF as an objective and quantitative assessment of neuromuscular block and its role in reducing postoperative complications has been demonstrated in numerous studies. In 2023, the "American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade" presented it with a moderate level of evidence and a high recommendation level. Likewise, in 2023, the European Society of Anesthesiology and Intensive Care's "Perioperative Management of Neuromuscular Blockade" guideline recommended TOF monitoring as part of routine perioperative monitoring with a 1B level of evidence .

TOF involves delivering four brief electrical impulses to a peripheral nerve at a frequency of 2 Hz and evaluating the resulting "twitches." The ratio of the response to the fourth stimulus to the response to the first stimulus (T4/T1) is referred to as the TOF ratio. Acceptable recovery of neuromuscular function is defined as a TOF ratio greater than or equal to 0.9. In a prospective study conducted in 2022 by Schmartz and colleagues, they compared a modified TOF ratio (T4/Tr) to the classic TOF ratio (T4/T1) against a reference measurement and demonstrated that the T4/Tr ratio is a better indicator of readiness for adequate recovery and safe extubation from non-depolarizing neuromuscular blockade compared to the classic TOF ratio (T4/T1) . This result suggests that the classic TOF ratio may overestimate the degree of true neuromuscular recovery, potentially leading to early tracheal extubation, increased risk of postoperative pulmonary complications, and endangering patient safety.

The aim of our study is to determine whether the differences in mTOF/classic TOF durations, as shown by Schmartz and colleagues in spontaneous neuromuscular recovery, also result in significant differences when rocuronium is reversed with sugammadex.

PROTOCOL:

Consent will be obtained from patients who meet the inclusion criteria during preoperative evaluation. After being admitted to the operating room, demographic information will be recorded and the following steps will be routinely performed.

Monitoring: ECG + NIKB + SpO2 + BIS + acceleromyography + body temperature Premedication: 1 mic/kg fentanyl and 0.05 mg/kg midazolam Preoxygenation: 3 minutes using 80% oxygen + 20% air with mask Anaesthesia Induction: 1 mic/kg fentanyl + 1 mg/kg lidocaine + 1 mg/kg propofol (BIS-guided) + 0.5 mic/kg breviblock Neuromuscular monitoring: After all standard preparations Set current to 50 mA Cancel T4/T2 TOF warning (1-2 times) 50 Hz tetanic stimulation for 5 s Calibration TOF warning until stabilisation is achieved (TOFr changes by less than 5% for 2-5 minutes) Muscle relaxation 1 mg/kg (according to ABW, actual) rocuronium/5 s bolus Analgesia 1 mic/kg fentanyl Intubation: Intubation with appropriately sized ETT when BIS is between 40-60, cTOFR: 0% Maintenance: BIS-guided TIVA anaesthesia (total 1 l/min oxygen and air mixture with FiO2 with SpO2 between 95-98) Muscle relaxant maintenance: PTC is measured at 5 minute intervals. PTC 1-2 is targeted. 5 mic/kg/min infusion is started. PTC measurement is continued. When PTC is 0, muscle relaxant infusion is stopped.

Intraoperative follow-up: PTC is measured at 5 minute intervals

* Stop rocuronium infusion if PTC is 0
* PTC 1-2 targeted values, 5 mic/kg/min maintenance rocuronium infusion is started.
* If PTC increases to 3 and above, 0.1 mg/kg bolus dose is added to the infusion. At the end of surgery : Anaesthetic drugs are switched off. PTC : 1-2, cTOFr measurement is started at 15 s intervals. 4 mg/kg sugammadex is administered. If cTOFR does not increase to 90% and above within 5 minutes, an additional dose of neostigmine is administered (0.02 mg/kg dose, without atropine).

Extubation: Extubation is performed when BIS is above 90% and cTOFR is 90% and above.

The patient is followed in the operating room until cTOFR and mTOFR are 100%.

During the perioperative course, the patient's TOFscan (cTOFR - mTOFR) data, the amount of neuromuscular blockers used, and the need for reversal medication are recorded.

STATISTICAL METHODOLOGY:

Sample Size The sample size required for the study was based on the difference between classical TOF and mTOF in neuromuscular recovery with Sugammadex. Accordingly, the required sample size for this study was calculated as 199 when the sample calculation was performed with the paired t test in dependent groups at 80% power and 0.05 significance level for a value of 0.2 indicating a low magnitude effect.

GPOWER 3.1 was used for sample calculation. Source: Cohen, J (1988). Statistical Power Analysis for the Social Sciences (2nd. Edition). Hillsdale, New Jersey, Lawrence Erlbaum Associates.

Statistical Methods Descriptive statistics will be given as frequency (%) for categorical variables, mean ± standard deviation and median (minimum-maximum) for continuous variables. In the comparison of dependent groups, paired t test will be used when the assumption of normal distribution is met and Wilcoxon test will be used when the assumption of normal distribution is not met. Statistical significance level will be accepted as p<0.05. The evaluation of the data will be done in SPSS 11.5 for Windows programme.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 (not including 65)
* BMI: 18.5-24.9

Exclusion Criteria:

* Liver and kidney disease
* Non-consenting
* Emergency surgeries
* Muscle disease
* Allergy to rocuronium and sugammadex
* Patients predicted to have difficult mask ventilation or difficult intubation
* Pregnant and breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgeries where neuromuscular blockers are used under general anesthesia
Sampling Method: Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
time | 15 minutes
  Comparison of classical and modified TOF rates to reach 90% and above

SECONDARY OUTCOMES:
time | 30 minutes
  Comparison of the time to reach 100% for classical and modified TOF rates

CONTACTS AND LOCATIONS:
Overall Officials: Menekşe Özçelik, 1, Study Director — Ankara University; Hatice Güneş Yeşilova, 2, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Altındağ, Turkey (Türkiye)

REFERENCES:
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Thilen SR, Weigel WA, Todd MM, Dutton RP, Lien CA, Grant SA, Szokol JW, Eriksson LI, Yaster M, Grant MD, Agarkar M, Marbella AM, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade: A Report by the American Society of Anesthesiologists Task Force on Neuromuscular Blockade. Anesthesiology. 2023 Jan 1;138(1):13-41. doi: 10.1097/ALN.0000000000004379. PMID 36520073
- [Background] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554
- [Background] Schmartz D, Bernard P, Sghaier R, Fils JF, Fuchs-Buder T. A modified TOF-ratio to assess rocuronium-induced neuromuscular block: a comparison with the usual TOF-ratio. Anaesth Crit Care Pain Med. 2022 Aug;41(4):101088. doi: 10.1016/j.accpm.2022.101088. Epub 2022 Apr 27. PMID 35489709